CLINICAL TRIAL: NCT05345119
Title: An Observational, Retrospective, Single-center, Clinical Study to Evaluate the Efficacy of Sirolimus (Rapamycin) in Patients With Graves' Disease and Moderate-to-severe and Active Graves' Orbitopathy (GO)
Brief Title: Sirolimus in Graves' Orbitopathy
Acronym: RETROSIRGO
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Associate Professor of Endocrinology, University of Pisa
Other Study IDs: RETROSIRGO
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Sirolimus; Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sirolimus: Treatment with sirolimus for 12 weeks, given as a second-line treatment
  Interventions: Drug: Sirolimus
- Methylprednisolone: Treatment with methylprednisolone for 12 weeks, given as a second-line treatment
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Sirolimus — 2 mg orally on the first day followed by 0.5 mg per day for 12 weeks
  Groups: Sirolimus
Drug: Methylprednisolone — 500 mg/weekly (6 weeks) intravenously, 250 mg/weekly (6 weeks) (cumulative dose 4.5 g).
  Groups: Methylprednisolone

SUMMARY:
Graves' Orbitopathy (GO) is a disabling and disfiguring condition associated with Graves' Disease, due to autoimmunity against antigens expressed by the thyroid and orbital tissues, and resulting in orbital fibroblast proliferation and release of glycosaminoglycans. The current treatments available, especially glucocorticoids, are not effective in all patients. Two cases of patients with GO treated with Sirolimus have been reported with an excellent response to the drug.

The rationale for the use of Sirolimus lies in its mechanisms of action. Sirolimus is able to inhibit T-cell activation as well as fibroblast proliferation. In addition, acts indirectly on the Insulin-Like Growth Factor-1 (IGF-1) pathway, and recent clinical trials have shown that a monoclonal antibody against the IGF-1 receptor (Teprotumumab) is effective in patients with GO. Thus, Sirolimus could be used in GO as monotherapy in patients with GO.

The aim of the present drug vs standard treatment, observational study is to evaluate the efficacy of Sirolimus as a second-line treatment in patients with moderately severe, active GO.

DETAILED DESCRIPTION:
Study Design: observational

Thirty consecutive patients with moderate-to-severe and active GO treated with sirolimus (15 patients) or methylprednisolone (15 patients) observance 18 consecutive months will be compared.

Study Timeline

Baseline visit - (Time 0) Treatment period (week 1-week 12): daily administration of the trial agent (Sirolimus) or weekly administration of the standard treatment (methylprednisolone) Outcome visit (week 24)

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
2. A moderate-to-severe GO, defined as the presence of at least one of the following criteria: an exophthalmos ≥2 mm compared with normal values for sex and race; presence of inconstant to constant diplopia; a lid retraction ≥2 mm
3. Active GO: CAS (4) ≥2 out of 7 points in the most affected eye
4. Previous GO treatment with glucocorticoids and/or orbital radiotherapy and/or orbital decompressive surgery, performed more than 24 weeks before the current treatment
5. Male and female patients of age: 18-75 years

Exclusion Criteria:

1. Optic neuropathy
2. Treatment with glucocorticoids or other immunosuppressive medications, and/or selenium, and/or orbital radiotherapy and/or orbital decompressive surgery in the 24 weeks preceding the current treatment
3. Mental illness that prevents patients from comprehensive, written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with moderate-to-severe, active Graves' orbitopathy treated with either sirolimus of methyprednisolone as a second-line treatment after a previous course of methyprednisolone, over 18 consecutive months
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
GO overall response | 24 weeks
  Percentage of subjects with at least two of the following compared to baseline: a) Improvement in clinical activity score (CAS) by at least 1 point ; b) Improvement in exophthalmos by at least 2 mm; c) Improvement in lid aperture by at least 2 mm; d) Improvement in eye muscle ductions ≥8 degrees; e) Improvement of visual acuity by at least 0.2/1, without worsening of any of these parameters in the contralateral eye if applicable.

SECONDARY OUTCOMES:
Change in exophthalmos | 24 weeks
  Percentage of subjects with a reduction greater than or equal to 2 mm compared with the baseline evaluation in the study eye, without worsening in the contralateral eye
Change in the clinical activity score (CAS) | 24 weeks
  Percentage of subjects with a reduction of CAS by at least two points in the study eye, without worsening in the contralateral eye
Change in quality of life | 24 weeks
  Comparison of the quality of life scores between the two groups, determined with a questionnaire specific for GO (GO-QoL)
Change in eye ductions | 24 weeks
  Percentage of subjects with an increase in eye ductions at least 8 degrees
Change in eyelid aperture | 24 weeks
  Percentage of subjects with a reduction greater than or equal to 2 mm
Change in diplopia | 24 weeks
  Percentage with an improvement in diplopia

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinologia II, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: Undecided